CLINICAL TRIAL: NCT00494078
Title: Efficiency of Real Time Continuous Glucose Monitoring to Achieve Normoglycemia in Critically Ill Patients - a Prospective, Randomized Study
Brief Title: Efficiency of Continuous Glucose Monitoring in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Ulrike Holzinger MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 488/2005
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2009-01

CONDITIONS: Critical Illness
Keywords: critical illness; hyperglycemia; intensive insulin therapy; glucose monitoring
MeSH Terms: conditions — Critical Illness; Hyperglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients randomised to this arm are treated with intensive insulin therapy guided by the continuous glucose monitoring system.
  Interventions: Device: Real-time glucose monitoring system (Guardian, Medtronic)
- 2 (Active Comparator): intensive insulin therapy guided by an algorithm
  Interventions: Drug: intensive insulin therapy

INTERVENTIONS:
Device: Real-time glucose monitoring system (Guardian, Medtronic) — Patients randomised to the intervention arm are treated with intensive insulin therapy guided by the real time glucose monitoring system.
  Other Names: Guardian (Medtronic); Novorapid (NovoNordisk)
  Arms: 1
Drug: intensive insulin therapy — intensive insulin therapy according to an algorithm
  Other Names: Novorapid (NovoNordisk)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether, real-time continuous glucose monitoring in critically ill patients with intensive insulin therapy would increase the percentage of time of normoglycemia, defined as glucose levels below 110 mg/dl.

DETAILED DESCRIPTION:
Hyperglycemia is associated with more complications and higher morbidity and mortality in critically ill patients. Therefore, strict glycemic control with a target blood glucose level between 80 and 110 mg/dl is recommended. Intensive insulin therapy requires continuous intravenous insulin infusion according to an algorithm and frequent blood glucose measurements. Implementation of intensive insulin therapy increases workload for both physicians and especially for nurses. The current gold-standard in intensive care units to achieve normoglycemia in critically ill patients is intensive insulin therapy according to a well established algorithm along with frequent blood glucose measurements. However, applying this gold-standard method, normoglycemia, defined as blood glucose levels below 110 mg/dl, can be achieved in approximately 50 percent of time only. We hypothesized, that real-time continuous glucose monitoring would increase the percentage of time of blood glucose levels below 110 mg/dl in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted critically ill patients expected to stay >48h on the ICU after initiation of intensive insulin therapy.
* Age > 18 years.

Exclusion Criteria:

* Admitted patients expected to stay <48h
* Age ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Percentage of time of normoglycemia, defined as glucose levels below 110 mg/dl, during the study period | 72h

SECONDARY OUTCOMES:
Median glucose levels during the study period; median time from start of intensive insulin therapy to achievement of normoglycemia; rate of hypoglycemias | 72h

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University of Vienna, Department of Medicine III
Locations (1):
- Medical University of Vienna, Vienna, Austria